CLINICAL TRIAL: NCT02515071
Title: Dietary Nitrate for OSAS: a Randomized, Placebo-controlled, Crossover Trial.
Brief Title: A 2 Week, Crossover Trial of Dietary Nitrate in Obstructive Sleep Apnoea Syndrome (OSAS).
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Royal College of Surgeons, Ireland (Other)
Collaborators: University College Dublin (Other); Connolly Hospital Blanchardstown (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: Chronic NO3- in OSAS
Record Dates: First submitted 2015-01-07; First posted 2015-08-04 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-08

CONDITIONS: Obstructive Sleep Apnoea Syndrome
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nitrate rich beetroot juice (Experimental): Concentrated, beetroot juice is a rich source of dietary nitrate.
  Interventions: Dietary Supplement: Dietary nitrate
- Nitrate depleted placebo beetroot juice (Placebo Comparator): Placebo beetroot juice is identical to active beetroot juice in every way except nitrate content.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Dietary nitrate — 140ml of nitrate rich beetroot juice provides 12.9mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Beetroot juice
  Arms: Nitrate rich beetroot juice
Dietary Supplement: Placebo — 140ml of nitrate depleted beetroot juice provides 0.5mmol nitrate and will be consumed on a daily basis during the intervention by the study subjects.
  Other Names: Nitrate depleted beetroot juice
  Arms: Nitrate depleted placebo beetroot juice

SUMMARY:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to decrease systemic blood pressure in multiple populations as well as increase organ perfusion in areas of interest such as the pancreas and brain. Obstructive sleep apnoea syndrome (OSAS) is associated with high blood pressure, dysglycaemia and impaired vigilance. The effect of dietary nitrate in OSAS has not been reported.

DETAILED DESCRIPTION:
Acute consumption of dietary nitrate (as beetroot juice) has been shown to decrease systemic blood pressure in multiple populations as well as increase organ perfusion in areas of interest such as the pancreas and brain. Obstructive sleep apnoea syndrome (OSAS) is associated with high blood pressure, dysglycaemia and impaired vigilance. The effect of dietary nitrate in OSAS has not been reported.

The investigators hypothesize that chronic nitrate consumption might decrease blood pressure and dysglycaemia and improve vigilance compared to a placebo beetroot juice.

This study is a randomized, double-blind placebo-controlled, crossover trial. At baseline, mid-point and endpoint ambulatory blood pressure will be assessed in conjunction with demographics, questionnaires, vigilance and blood draw. After baseline measures, each subject will be randomized to consume nitrate rich beetroot juice for 14 consecutive nights when assessments will be repeated followed by 14 nights of placebo and endpoint assessments or the converse.

ELIGIBILITY:
Inclusion Criteria:

* Clinically stable,
* Untreated OSAS out-patients

Exclusion Criteria:

* Using continuous positive airways pressure therapy
* Pulmonary hypertension
* Active CVD
* Active musculo-skeletal conditions
* Taking vasodilators
* Diabetes mellitus

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Difference in ambulatory nocturnal blood pressure | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.

SECONDARY OUTCOMES:
Difference in 24h blood pressure | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in plasma nitrate and nitrite | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in fasting glucose | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in OSAS symptomatology | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in 2h post OGT glucose | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in overnight oximetry | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in exhaled nitric oxide | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.
Difference in vigilance scores derived from the Conner's Continuous Performance Test. | Day 1, day 15, day 29
  Comparison of the change after nitrate-rich beetroot juice compared to placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Liam Cormican, MD, Principal Investigator — Connolly Hospital
Locations (1):
- Connolly Hospital, Blanchardstown, Dublin, Ireland